CLINICAL TRIAL: NCT03076047
Title: Preliminary Characterization of the Capnography Profile of Obstructive Sleep Apnea (OSA) Patients in the Post-Anesthesia Care Unit (PACU)
Brief Title: Capnography in the Post-Anesthesia Care Unit (PACU)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Principal Investigator, Enrico Camporesi, Principal Investigator, University of South Florida
Other Study IDs: Pro00027304
Record Dates: First submitted 2017-03-06; First posted 2017-03-09 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Obstructive Sleep Apnea; Bariatric Surgery Candidate; Respiratory Insufficiency
MeSH Terms: conditions — Sleep Apnea, Obstructive; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- end tidal CO2 (ETCO2) monitoring: We will continuously record capnography data from the patients while they are in the post-anesthesia care unit (PACU). Study personnel will visit each patient while the patient is in the PACU to promote compliance with continuous CO2 monitoring.
  Interventions: Device: end-tidal CO2 (ETCO2) monitoring

INTERVENTIONS:
Device: end-tidal CO2 (ETCO2) monitoring — monitor end tidal CO2 levels while patients recover in post-anesthesia care unit (PACU) using the Smart CapnoLine Plus O2, Capnostream, and Massimo

SUMMARY:
To understand if a progressive increase in end-tidal carbon dioxide (CO2) levels are heralding respiratory difficulties before desaturation measured from capnography in obstructive sleep apnea patients, with the use of nasal prongs, transcutaneous monitors, Capnostream, and Massimo technologies.

DETAILED DESCRIPTION:
Background and Significance Carbon dioxide (CO2) levels can be monitored throughout the respiratory cycle via capnography. In this way, capnography allows healthcare professionals to follow a number of respiratory factors (i.e., depression, apnea, and hypercapnia) in real-time. Earlier detection of alterations to ventilation status will better enable providers to more accurately dose medications during procedures, especially in at-risk patient populations such as patients with obstructive sleep apnea (OSA) [1, 2].

In a recent study of bariatric patients, approximately 15% experience postoperative pulmonary complications. These patients could benefit significantly from capnography monitoring as this measure can very accurately estimate the prevalence of respiratory complications.

Through this study we seek to understand how end-tidal CO2 (ETCO2) levels of patients with obstructive sleep apnea vary when patients are in the post-anesthesia care unit (PACU). By collecting information on patient outcomes, we hope to better understand the value of this monitoring technique in an at-risk patient population. Though capnography in the PACU has not previously been demonstrated to improve patient safety or satisfaction, capnography has never been studied in a population of patients who are at risk of obstructive sleep apnea.

Study Design This is a prospective, blinded observational pilot study to monitor if changes in end-tidal CO2 levels provide incremental value over pulse oximetry when detecting respiratory difficulties (i.e., hypercapnia).

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Patients who have are at TGH for bariatric surgery
* BMI > 30
* At risk of obstructive sleep apnea according to TGH STOP-BANG questionnaire

Exclusion Criteria:

* <18 years of age
* Not at risk of obstructive sleep apnea according to TGH STOP-BANG questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at high-risk of obstructive sleep apnea undergoing gastric bypass surgery
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2023-02-09 (Estimated); Study Completion 2023-02-09 (Estimated)

PRIMARY OUTCOMES:
end-tidal carbon dioxide (ETCO2) | 2-3 hours
  end-tidal carbon dioxide (ETCO2) values averaged over 5 minute intervals

SECONDARY OUTCOMES:
oxygen saturation (SPO2) | 2-3 hours
  oxygen saturation (SPO2) values from pulse oximetry

CONTACTS AND LOCATIONS:
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta PP, Kochhar G, Albeldawi M, Kirsh B, Rizk M, Putka B, John B, Wang Y, Breslaw N, Lopez R, Vargo JJ. Capnographic Monitoring in Routine EGD and Colonoscopy With Moderate Sedation: A Prospective, Randomized, Controlled Trial. Am J Gastroenterol. 2016 Mar;111(3):395-404. doi: 10.1038/ajg.2015.437. Epub 2016 Feb 23. PMID 26902229
- [Background] Barnett S, Hung A, Tsao R, Sheehan J, Bukoye B, Sheth SG, Leffler DA. Capnographic Monitoring of Moderate Sedation During Low-Risk Screening Colonoscopy Does Not Improve Safety or Patient Satisfaction: A Prospective Cohort Study. Am J Gastroenterol. 2016 Mar;111(3):388-94. doi: 10.1038/ajg.2016.2. Epub 2016 Feb 2. PMID 26832654